CLINICAL TRIAL: NCT05218681
Title: Measuring and Reducing Substance Use Disorder Stigma Among Hospital-based Nurses
Brief Title: Nursing Attitudes Towards SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 849369
Record Dates: First submitted 2021-11-15; First posted 2022-02-01 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Substance Use Disorders; Stigma, Social
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Unit-based "Person First" Anti-stigma Awareness Rounds (Other): The "Person First" Initiative was developed independent of this study by bedside nurses (including McFadden) in collaboration with HUP Nursing Executive Leadership. The objective of this initiative is to provide (1) unit-based "huddles" on person-first language as a mechanism to reduce the stigma around substance use; (2) socialize best practices and resources for patients with substance use disorder; and (3) provide overdose reversal training and kits, including Narcan nasal spray, to nurses. The planning and implementation of these activities fall under the purview of Nursing Shared Governance (NOT the research team), and oversight for these activities will be provided by HUP Nursing Executive Leadership.
  Interventions: Other: Unit-based "Person First" Anti-stigma Awareness Rounds
- Unit-based "Person First" stigma rounds + Text-based Messaging (Other): Participating nurses will be randomized to receive weekly short text messages that employ evidence-based strategies to reduce stigma towards individuals with substance use disorder over the course of 6-months.
  Interventions: Other: Unit-based "Person First" Anti-stigma Awareness Rounds; Other: Individual Text-based Messaging

INTERVENTIONS:
Other: Unit-based "Person First" Anti-stigma Awareness Rounds — Educational rounds on stigma
Other: Individual Text-based Messaging — Weekly evidence based messages to reduce SUD stigma
  Arms: Unit-based "Person First" stigma rounds + Text-based Messaging

SUMMARY:
The purpose is to measure substance use disorder (SUD)-related stigma among hospital-based nurses using validated survey instruments, and attempt to reduce stigma through a combination of individual and unit-based educational and participatory interventions.

DETAILED DESCRIPTION:
The proposed research is a pre-/post-survey, qualitative study of substance use disorder-related stigma among nurses and a sustained, "bundled" intervention to reduce this stigma. The objectives of the study are to:

1. Measure existing substance use disorder (SUD) stigma among nurses at HUP;
2. Evaluate the effects of combined individual and unit-based stigma-reduction interventions; and
3. Adapt and psychometrically analyze a stigma assessment instrument tailored to hospital-based health care providers.

The study team will approach unit-based nursing leadership on target units regarding participation in the (1) unit-based education/awareness activities and (2) individual-based survey and randomized intervention. The study team may meet virtually with unit-based nursing leadership, and/or present the intervention and survey opportunity during unit council meetings per the request of leadership. The study team will send an email to the complete unit nursing listserv. The email from the study team will contain information about the study, contact information, and consent form. Once the ICF has been electronically signed by a participant, the Way to Health platform will generate and send an electronic message to the participant containing a link to the survey.

After 6-months , nurses who completed the ICF & pre-survey previously will receive electronic prompts from Way to Health to complete the post-survey. The survey will first be made available to pre-survey completers. After 2 weeks, the survey opportunity will be opened to non-enrolled nurses on the participating unit; this will be communicated to the participating unit by the study team via an email to the nursing listserv, which will includeThe email from the study team will contain information about the study, contact information, and consent form. The ICF must be electronically signed by a participant in order for the survey to become available.

Interventions:

1. Unit-based "Person First" Anti-stigma Awareness Rounds The "Person First" Initiative was developed independent of this study by bedside nurses in collaboration with HUP Nursing Executive Leadership. The objective of this initiative is to provide (1) unit-based "huddles" on person-first language as a mechanism to reduce the stigma around substance use; (2) socialize best practices and resources for patients with substance use disorder; and (3) provide overdose reversal training and kits, including Narcan nasal spray, to nurses. The planning and implementation of these activities fall under the purview of Nursing Shared Governance (NOT the research team), and oversight for these activities will be provided by HUP Nursing Executive Leadership (Chief Nursing Executive Colleen Mattioni and Director of Ethics Aliza Narva). The goal of the "Person First" initiative is to engage with every unit at HUP, although level of engagement (e.g. single round vs multiple rounds) will vary by unit capacity and interest, and some units may opt out of these activities.
2. Individual Text-based Messaging Participating nurses will be randomized to (1) receive short text messages that employ evidence-based strategies to reduce stigma towards individuals with substance use disorder, or (2) no messaging. Pre-determined messages will be sent via Way to Health weekly for 6 months to the phone number provided by participants during the consent process. Participants will have the option to stop receiving these messages at any time.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses working in any capacity (bedside, administration) at the Hospital of the University of Pennsylvania.

Exclusion Criteria:

* If a nursing leadership on a unit declines survey participation for their unit, nurses who work on that unit will not be recruited/included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change in stigma towards patients with Substance use disorder on the individual nursing level | 6-months
  Change in stigma towards patients with substance use disorder based on pre-post survey among individual nurses. Nurses will be given the same survey pre and post-intervention. The survey includes a Modified stigma score where likert scales are dichotomized as follows:
  * Very Approriate, Appropriate vs Other
  * Strongly agree and agree vs other

SECONDARY OUTCOMES:
Change in stigma on the unit-level | 6-months
  Change in stigma towards patients with substance use disorder based on pre-post survey across units. Nurses will be given the same survey pre and post-intervention. The survey includes a Modified stigma score where likert scales are dichotomized as follows:
  * Very Approriate, Appropriate vs Other
  * Strongly agree and agree vs other

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided